CLINICAL TRIAL: NCT06785350
Title: Minimum Effective Dose of Incisional Local Infiltration Betamethasone for the Prevention of Pain After Spinal Surgery: a Randomised Controlled Trial
Brief Title: Minimum Effective Dose of Incisional Local Infiltration Betamethasone for the Prevention of Pain After Spinal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Tiantan Hospital (Other)
Responsible Party: Principal Investigator, Fang Luo, Director of Department of Pain Management, Beijing Tiantan Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: KY2024-365-02-1
Record Dates: First submitted 2025-01-04; First posted 2025-01-21 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Pain Management; Spine Surgery
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- intervention group 1 (Experimental): 0.012%diprospan+0.5%ropivacaine
  Interventions: Drug: 0.012%diprospan+0.5%ropivacaine
- intervention group 2 (Experimental): 0.009%diprospan+0.5%ropivacaine
  Interventions: Drug: 0.009%diprospan+0.5%ropivacaine
- intervention group 3 (Experimental): 0.006%diprospan+0.5%ropivacaine
  Interventions: Drug: 0.006%diprospan+0.5ropivacaine
- intervention group 4 (Experimental): 0.003%diprospan+0.5%ropivacaine
  Interventions: Drug: 0.003%diprospan+0.5%ropivacaine
- control group (Active Comparator): 0.5%ropivacaine
  Interventions: Drug: 0.5%ropivacaine

INTERVENTIONS:
Drug: 0.012%diprospan+0.5%ropivacaine — At the preoperative visit, patients will sign informed consent and learn to use the patient-controlled analgesia (PCA) pump and assess pain with the visual analogue scale (VAS). Standard general anesthesia will be induced and maintained with sufentanil, propofol, cisatracurium or rocuronium, and sevoflurane. Before incision, neurosurgeons will administer the allocated local infiltration solution. 0.5ml of diprospan will be diluted to 30 ml with 15 ml of ropivacaine in 0.9% NaCl to prepare diprospan at concentrations of 0.012%, respectively. The surgeon will use a 22 G straight needle for local infiltration anesthesia near the planned incisions. Postoperatively, patients will receive tropisetron and a PCA pump delivering sufentanil and ondansetron. PCA usage (effective/ineffective presses) and supplemental analgesia with Tylenol or loxoprofen will be monitored for 48 hours and up to 3 months. Dosages and intraoperative parameters will be closely recorded throughout.
  Arms: intervention group 1
Drug: 0.009%diprospan+0.5%ropivacaine — At the preoperative visit, patients will sign informed consent and learn to use the patient-controlled analgesia (PCA) pump and assess pain with the visual analogue scale (VAS). Standard general anesthesia will be induced and maintained with sufentanil, propofol, cisatracurium or rocuronium, and sevoflurane. Before incision, neurosurgeons will administer the allocated local infiltration solution. 0.375ml of diprospan will be diluted to 30 ml with 15 ml of ropivacaine in 0.9% NaCl to prepare diprospan at concentrations of 0.009%, respectively. The surgeon will use a 22 G straight needle for local infiltration anesthesia near the planned incisions. Postoperatively, patients will receive tropisetron and a PCA pump delivering sufentanil and ondansetron. PCA usage (effective/ineffective presses) and supplemental analgesia with Tylenol or loxoprofen will be monitored for 48 hours and up to 3 months. Dosages and intraoperative parameters will be closely recorded throughout.
  Arms: intervention group 2
Drug: 0.006%diprospan+0.5ropivacaine — At the preoperative visit, patients will sign informed consent and learn to use the patient-controlled analgesia (PCA) pump and assess pain with the visual analogue scale (VAS). Standard general anesthesia will be induced and maintained with sufentanil, propofol, cisatracurium or rocuronium, and sevoflurane. Before incision, neurosurgeons will administer the allocated local infiltration solution. 0.25ml of diprospan will be diluted to 30 ml with 15 ml of ropivacaine in 0.9% NaCl to prepare diprospan at concentrations of 0.006%, respectively. The surgeon will use a 22 G straight needle for local infiltration anesthesia near the planned incisions. Postoperatively, patients will receive tropisetron and a PCA pump delivering sufentanil and ondansetron. PCA usage (effective/ineffective presses) and supplemental analgesia with Tylenol or loxoprofen will be monitored for 48 hours and up to 3 months. Dosages and intraoperative parameters will be closely recorded throughout.
  Arms: intervention group 3
Drug: 0.003%diprospan+0.5%ropivacaine — At the preoperative visit, patients will sign informed consent and learn to use the patient-controlled analgesia (PCA) pump and assess pain with the visual analogue scale (VAS). Standard general anesthesia will be induced and maintained with sufentanil, propofol, cisatracurium or rocuronium, and sevoflurane. Before incision, neurosurgeons will administer the allocated local infiltration solution. 0.125ml of diprospan will be diluted to 30 ml with 15 ml of ropivacaine in 0.9% NaCl to prepare diprospan at concentrations of 0.003%, respectively. The surgeon will use a 22 G straight needle for local infiltration anesthesia near the planned incisions. Postoperatively, patients will receive tropisetron and a PCA pump delivering sufentanil and ondansetron. PCA usage (effective/ineffective presses) and supplemental analgesia with Tylenol or loxoprofen will be monitored for 48 hours and up to 3 months. Dosages and intraoperative parameters will be closely recorded throughout.
  Arms: intervention group 4
Drug: 0.5%ropivacaine — At the preoperative visit, patients will sign informed consent and learn to use the patient-controlled analgesia (PCA) pump and assess pain with the visual analogue scale (VAS). Standard general anesthesia will be induced and maintained with sufentanil, propofol, cisatracurium or rocuronium, and sevoflurane. Before incision, neurosurgeons will administer the allocated local infiltration solution. 15 ml of ropivacaine will be diluted to 30 ml with in 0.9% NaCl, respectively. The surgeon will use a 22 G straight needle for local infiltration anesthesia near the planned incisions. Postoperatively, patients will receive tropisetron and a PCA pump delivering sufentanil and ondansetron. PCA usage (effective/ineffective presses) and supplemental analgesia with Tylenol or loxoprofen will be monitored for 48 hours and up to 3 months. Dosages and intraoperative parameters will be closely recorded throughout.
  Arms: control group

SUMMARY:
Incisional pain is a common complication after surgery and is an important cause of delayed postoperative recovery, increased length of hospital stay, increased risk of wound infection and respiratory/cardiovascular complications, as well as an important medical, social, and economic problem. Prevention and treatment of postoperative incision pain remains challenging. Local Infiltration Anaesthesia (LIA) for surgical incisions with an anti-inflammatory and analgesic combination has been reported to be effective in reducing postoperative pain, but there is a gap in the research on the optimal concentration of anti-inflammatory drugs in the anti-inflammatory and analgesic combination during local infiltration. The aim of this study was to investigate the optimal concentration of anti-inflammatory drugs in the anti-inflammatory-analgesic combination solution used for local infiltration of spinal surgical incisions to prevent postoperative pain.

ELIGIBILITY:
Inclusion Criteria:

Patients scheduled for spine surgery under general anesthesia. Anticipated cervical, thoracic, and lumbar spine surgeries (within three level).

Patients age 18-65 years. American Society of Anaesthesiologists Classification of I or II.

Exclusion Criteria:

Patients refuse to participate. Patients who are allergic to ropivacaine, betamethasone and opioid, . Pateints who have been abusing drugs or alcohol. Patients who have abnormalities in kidney or liver function tests. BMI<15kg/m2 or>35 kg/m2. Patient has a history of spinal surgery. Patient has peri-incisional infection. Patient has a history of stroke or other serious neurological disease. Patient has a history of diabetes and other metabolic disorders. Patient has a history of psychological disorders. Patient is on systemic steroids. Patient is pregnant or breastfeeding. Glasgow Coma Scale score < 15 before surgery. Unable to provide written informed consent.

Withdrawal criteria:

Voluntary withdrawal. Delayed extubation. Poor cognitive function within 48 hours after surgery. Postoperative radiation therapy or chemotherapy during follow-up. Postoperative diagnosis of spinal cord or nerve root injury resulting in pain during follow-up.

Reoperation during follow-up.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 535 (Estimated)
Dates: Start 2025-01-25 (Actual); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
postoperative sufentanil consumption via PCA | At 48 hours after the operation
  The cumulative 48 hours postoperative sufentanil consumption via PCA was the primary outcome of our study

SECONDARY OUTCOMES:
Cumulative consumption of sufentanil by PCA | During 0-4hours, 4-8hours, 8-24hours and 24-48hours after operation
PCA pump first press time | Within 48 hours after the operation.
VAS score at during movement (VASm) and at rest (VASr) | At 2hours, 4hours, 8hours, 24hours, 48hours, 72hours, 1week, 2weeks, 6weeks, 3months postoperatively
  0 indicates no pain, 10 indicates the most severe pain imaginable.
Intraoperative opioid dosage | During the operation
Time to first analgesic remediation | Until 3 months after surgery
Amount of postoperative oral analgesic remediation | Until 3 months after surgery
Postoperative nausea and vomiting (POVN) | At 2hours, 4hours, 8hours, 24hours, and 48hours postoperatively
  PONV will be rated by participants as: 0, absent; 1, nausea not requiring treatment; 2, nausea requiring treatment; and 3, vomiting.
Ramsay sedation score (RSS) | At 2hours, 4hours, 8hours, 24hours, 48hours postoperatively
  Ramsey 1: Anxious, agitated, restless; Ramsey 2: Cooperative, oriented, tranquil; Ramsey 3: Responsive to commands only If Asleep; Ramsey 4: Brisk response to light glabellar tap or loud auditory stimulus; Ramsey 5: Sluggish response to light glabellar tap or loud auditory stimulus; Ramsey 6: No response to light glabellar tap or loud auditory stimulus.
Satisfaction score | At 2hours, 4hours, 8hours, 24hours, 48hours, 72hours, 1week, 2weeks, 6weeks, 3months postoperatively
  0 for unsatisfactory, and 10 for very satisfied
The World Health Organization Quality of Life (WHOQOL) | At 3months postoperatively
  Higher scores indicate a better perception of quality of life.
Oswestry disability index (ODI) | At 3months postoperatively
  The Oswestry Disability Index (ODI) is a widely used tool to measure disability related to lower back pain. It consists of 10 sections, each addressing different aspects of daily life affected by back pain. Higher scores mean more severe pain.
Patient and Observer Scar Assessment Scale (POSAS) | At 3months postoperatively
  The Patient and Observer Scar Assessment Scale (POSAS) is a widely used tool for assessing scars from both the patient's and observer's perspectives. It evaluates scar quality based on physical characteristics and the patient's subjective experience. Lower scores indicate better scar quality and fewer issues. Higher scores reflect worse scar quality or greater subjective dissatisfaction.
Adverse events | At 3months postoperatively

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in this article, after de-identification (text, tables, figures and appendices) are available. Derived data supporting the findings of this study are available from the corresponding author Fang Luo on request.

REFERENCES:
- [Derived] Wang Y, Han B, Zhao C, Ren H, Jia W, Luo F. Minimum effective dose of betamethasone for incisional local infiltration for the prevention of postoperative pain after spine surgery: study protocol for a randomised controlled trial. BMJ Open. 2025 Sep 28;15(9):e100725. doi: 10.1136/bmjopen-2025-100725. PMID 41022457